CLINICAL TRIAL: NCT02681627
Title: Pilot Randomised Controlled Trial of the Effect of Endometrial Scratch in Recurrent Miscarriage on Pregnancy Outcomes
Brief Title: Sim (Scratch in Miscarriage) Study
Acronym: SiM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Rego2015 1630
Record Dates: First submitted 2016-02-03; First posted 2016-02-12 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Miscarriage
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- endometrial scratch (Active Comparator): Patient will be randomised to the intervention arm which is the luteal phase endometrial scratch
  Interventions: Other: Endometrial scratch
- touching cervix (Sham Comparator): Patient will have a speculum examination and cleaning of the cervix with cotton tip with saline but no scratch
  Interventions: Other: Touching the cervix

INTERVENTIONS:
Other: Endometrial scratch — If patient randomised to intervention arm, will have speculum examination followed by endometrial scratch with a wallace catheter
  Arms: endometrial scratch
Other: Touching the cervix — If patient is randomised to the control arm, she will have speculum examination followed by cleaning of the cervix with a cotton tip dipped in saline
  Arms: touching cervix

SUMMARY:
There is increasing amount of evidence which suggests that miscarriage is related to a primary endometrial problem. Recent cochrane meta-analysis (March 2015) has proven that endometrial scratch improves live birth in women who underwent IVF.

The aim of the study is to find out if scratch of the endometrium prevents recurrent miscarriage.

DETAILED DESCRIPTION:
The Warwick BRU-RH (Biomedical Research Unit- Reproductive Health) hypothesis is that failed pregnancies are the result of failed decidualisation of the endometrium.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Actively trying for a pregnancy

Exclusion Criteria:

1. No active treatment in pregnancy
2. Inherited or acquired thrombophilia
3. Medical conditions- diabetes,hypertension,thyroid disorders
4. inability to tolerate internal examinations
5. uterine anomalies
6. Previous entry or randomisation in the present trial

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate after 24 weeks of gestation | from the recruitment of the first patient up to 12 months after the recruitment of last patient. the live birth rate of all the pregnant patients in the study who delivered after 24 weeks will be included in the outcome.

SECONDARY OUTCOMES:
Miscarriage until 23+6 weeks of gestation | from the recruitment of the first patient and up to 12 months after the recruitment of last patient. the outcomes of all the pregnant patients in the study who delivered up to 23+6 weeks will be included in the outcome.
Pregnancy complications | from the recruitment of the first patient and up to 12 months after the recruitment of last patient. The patients who delivered after 24 weeks with a live birth will be included in the outcome and the described outcomes will be measured
  Such as SGA(small for gestational age),PET( Pre-eclamptic toxaemia),Abruption, Placenta Praevia, Placenta accreta and Preterm delivery
Acceptability of the intervention | Patient questionnaire will be issued at the time of randomisation. the returned forms up to 4 weeks after randomisation will be analysed and reported. this will be helpful for assessing the patients tolerability of the procedure
  To guide future trial set up

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Quenby, MD FRCOG, Principal Investigator — UHCW NHS Trust
Locations (1):
- University Hospitals of Coventry and Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom